CLINICAL TRIAL: NCT01322178
Title: Open-label, Uncontrolled, Multi-center, Phase II Study of Cetuximab in Combination With mFOLFOX-6 as First-line Treatment in Patients With KRAS Wild-type, Unresectable LIver Metastases of colorEctal Cancer
Brief Title: Study of Cetuximab in Combination With mFOLFOX-6 (Oxaliplatin, Leucovorin, 5-FU) to Treat Colorectal Liver Metastatic Cancer Patients
Acronym: CLIME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sanjun Cai, Fudan University Shanghai Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-203
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: cetuximab; colorectal carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cetuximab; mFOLFOX6 — Cetuximab (Erbitux): 500 mg/m2 iv gtt, D1
  Oxaliplatin: 85 mg/m2 iv gtt over 2 hours, D1; leucovorin: 400 mg/m2 iv gtt , D1; 5-FU: 400 mg/m2 iv, 2400 mg/m2 civ46h
  repeated every two weeks for 4.5 months(9 cycles)

SUMMARY:
The aim of this study is to explore whether cetuximab in combination with mFOLFOX6 as treatment could improve the resection rate in patients with KRAS wild-type, unresectable liver metastases of mCRC.

DETAILED DESCRIPTION:
During the last decade, chemotherapy in metastatic colorectal cancer (mCRC) has made considerable progress.However, approximately 25% of patients with colorectal cancer present with overt metastatic disease. In selected patients, synchronous or metachronous liver metastases (LM) can be resected in curative intention. Over the last 5 years there has been the recognition that preoperative, neoadjuvant, combination chemotherapy regimens, namely, 5-fluorouracil/folinic acid (5-FU/FA) in combination with either irinotecan or oxaliplatin can facilitate to downsize the initially unresectable LM and make the resection possible. The addition of targeted therapies might render them even more effective.

Due to these results, the investigators hypothesize that cetuximab in combination with mFOLFOX6 as treatment in patients with KRAS wild-type, unresectable liver metastases of mCRC may further improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-75 years of age
* Performance status (ECOG) 0~1
* Unresectable, histologically confirmed, synchronous or metachronous liver metastasis of colorectal cancer. Unresectable liver metastases is defined as:

  * patients with five and more liver metastases and/or
  * Liver metastases that are technically unresectable immediately, and expected remaining functional liver tissue ≥ 30% after resection. (Patients should be evaluated by a multidisciplinary team of three local surgeons and one local radiologist, including surgical consultation for potentially resectable patients on the basis of remaining liver volume, infiltration of all liver veins, infiltration of both liver arteries, both portal branches or both bile ducts.)
* Tumor tissue (primary or metastasis) genotypologically classified as KRAS wild-type in codon 12 and codon 13 of the KRAS gene exon 2
* No prior chemotherapy (except adjuvant chemotherapy with an interval of ≥ 6 months)
* Presence of at least one index lesion of hepatic metastasis measurable by CT scan or MRI, not in an irradiated area
* Neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 8 g/dL
* Bilirubin level ≤ 1.0 x ULN
* AST and ALT < 1.5 x ULN
* Serum creatinine ≤ 1.0 x ULN
* Life expectancy of ≥ 3 months
* Male or female of child-bearing period should have effective contraception
* Signed written informed consent

Exclusion Criteria:

* Any investigational agent(s) within 4 weeks prior to entry
* Previous exposure to EGFR-targeting therapy
* Any evidence of extrahepatic metastases and/or primary tumor recurrence
* Total volumes of liver lesions > 70%
* Clinically relevant peripheral neuropathy
* Acute or sub-acute intestinal obstruction or history of inflammatory bowel disease
* Breast-feeding or pregnant women, no effective contraception if risk of conception exists (for male and female patients up to 4 months after end of chemotherapy)
* Previous malignancy (except colorectal cancer, history of basal cell carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment)
* Known drug abuse/ alcohol abuse
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Severe organ failures or diseases, including: clinically relevant coronary disease, cardiovascular disorder or myocardial infarction within 12 months before study entry, severe psychiatric illness, severe infection and DIC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Resection rate (R0) | from the first cycle of treatment (day one) to two month after the last cycle

SECONDARY OUTCOMES:
Response rate,Progression-free Survival,Overall Survival,R1 resection rate | from the first cycle of treatment (day one) to six month after the last cycle
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | from the first cycle of treatment (day one) to six month after the last cycle

CONTACTS AND LOCATIONS:
Overall Officials: Sanjun Cai, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China